CLINICAL TRIAL: NCT02624895
Title: ProSpective multIcenter observationaL Study on the Quality of Life of mCRC RAS Wild-type Patients Receiving Anti-EGFR MAbs + FOLFOX or FOLFIRI as 1st Line of Treatment
Brief Title: ObservationaL Study on the Qol of RAS Wild-type mCRC Patients Receiving Anti-EGFR MAbs + FOLFOX or FOLFIRI as 1st Line
Acronym: SILQ
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140383
Record Dates: First submitted 2015-11-09; First posted 2015-12-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer gene RAS not mutated "WILD TYPE"
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — not collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mCRC: Anti-EGFR MAbs + FOLFOX 1st line: • Adult (>= 18 years old) RAS wild-type metastatic colorectal cancer patients candidate to receive FOLFOX plus panitumumab or FOLFOX plus cetuximab as upfront treatment as per clinical practice.
- mCRC: Anti EGFR MAbs + FOLFIRI 1st line: Adults (>= 18 years old) RAS wild-type metastatic colorectal cancer patients candidate to receive FOLFIRI plus panitumumab or FOLFIRI plus cetuximab as upfront treatment as per clinical practice

SUMMARY:
This is a national, multicentric, prospective, observational trial. The decision to prescribe FOLFOX or FOLFIRI plus panitumumab or FOLFOX or FOLFIRI plus cetuximab must have been freely taken by the clinician prior to the study entry for each patient included. Each physician will see his/her patients within the context of routine visits, without any special visit being organised for the purposes of the study. Therefore, the doctor-patient relationship and patient follow-up are not modified. Physicians are totally free to decide on their patients' therapeutic management.

EORTC QLQ-C30 and DLQI questionnaires will be completed by the patients at baseline (Day 1 of Cycle 1), at the first day of every other cycle (every 2 weeks) thereafter, and at ""End of Study Visit" (within 28 days from the end of treatment with anti-EGFR or withdrawal from study for any reason).

Before every cycle, adverse events will be recorded and graded according to NCI CTCAE v4.0. Treatment's modifications in terms of cycles' delay, dose reductions or drugs' interruptions will be recorded.

Concomitant approaches to prevent or treat dermatological toxicities during the treatment will be registered.

ELIGIBILITY:
Inclusion Criteria:- Adult (>= 18 years old) RAS wild-type metastatic colorectal cancer patients candidate to receive FOLFOX or FOLFIRI plus panitumumab or FOLFOX or FOLFIRI plus cetuximab as upfront treatment as per clinical practice

* Willingness and ability to comply with the protocol
* Written informed consent to study procedures
* Exclusion Criteria: - Patients receiving a treatment under clinical investigation may not be included in the study
* Previous treatment with an anti-EGFR monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>= 18 years old) RAS wild-type metastatic colorectal cancer patients candidate to receive FOLFOX or FOLFIRI plus panitumumab or FOLFOX or FOLFIRI plus cetuximab as upfront treatment as per clinical practice. Willingness and ability to comply with the protocol. Written informed consent to study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ C30 questionnaire score | 24 months
  -HRQoL will be measured using the EORTC QLQ-C30 questionnaire. EORTC QLQ-C30 scores reported during the treatment will be also expressed as percentage of the scores reported at baseline. The measure unit is the answer score provided by the patient to the questions in the questionnaire
QoL questionnaire DLQI questionnaire score | 24 months
  Skin satisfaction will be measured using the DLQI. The DLQI score will also be expressed as a percentage of the maximum possible score of 30. DLQI scores reported during the treatment will be also expressed as percentage of the DLQI scores reported at baseline.The measure unit is the answer score provided by the patient to the questions in the questionnaire
%of enrolled subjects, experiencing a specific adverse event according to NCI CTC-AE version 4.0 | 24 months
  Tolerability: The toxicity rate, defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of any grade, according to CTCAE version 4.02.
Recording of number of concomitant medications, to prevent or treat dermatological adverse events | 24 months
  Management of dermatological toxicity: concomitant medications, both topical and systemic, adopted to prevent or treat dermatological adverse events will be recorded. The measure is the number of topical and systemic treatment administered for skin toxicity management
Time to onset of the dermtological toxicity | 24 months
  Tolerability: Times to onset of dermatological toxicities will be also described. The measure is the times elapsed untill adverse event is occurred (days)
Dose reduction | 24 months
  To describe the adherence to the treatment in terms of dose reduction.The measure unit is Number of dose reduction occurred out of standard as per clinical practice treatment scheme.
"number of administered cycles" | 24 months
  Evaluate the number of treatment cycles performed by the patients. The measure is the number of cycles administered as per clinical practice scheme indicated in the protocol, by each patient
average relative dose intensity of every drug" | 24 months
  Will be evaluated the average dose administered to the patient under treatment the measure units are mg or mg/kg

SECONDARY OUTCOMES:
Score scale on questionnaire answers | 24 months
  To investigate the impact of dermatological adverse events during the treatment with FOLFOX plus anti-EGFR MAbs on patients' skin satisfaction as measured by means of the Dermatology Life Quality Index (DLQI) questionnaire. The measure unit is the score coming from patient answer to questions in the questionnaire
Number of cycles on treatment before and of treatment due to AE | 24 months
  To assess the tolerability of administered treatments The measure unit is the number of cycles on treatment before and of treatment due to AE
dose delay | 24 months
  To describe the adherence to the treatment in terms of dose delays, - the measure unit is Number of dose delay occurred out of standard as per clinical practice treatment scheme
Questionnaire score | 24 months
  To describe the management of dermatological adverse events to assess the effect on skin-related QoL of preemptive Vs reactive treatment of skin toxicities. The measure units is the questionnaire score coming from patient answer to relevant questionnaire administered.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (28):
- Italy (28):
  - Research Site, Brescia
  - Research Site, Castellana Grotte
  - Research Site, Castellanza (VA)
  - Research Site, Catania
  - Research Site, Cona FE
  - Research Site, Confreria - Cuneo
  - Research Site, Crema
  - Research Site, Fano PU
  - Research Site, Foggia
  - Research Site, Frattamaggiore NA
  - Research Site, Isernia
  - Research Site, Lecce
  - Research Site, L’Aquila
  - Research Site, Mirano VE
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Poggibonsi SI
  - Research Site, Potenza
  - Research Site, Rionero in Vulture (PZ)
  - Research Site, Roma
  - Research Site, Roma (RM)
  - Research Site, Sanremo (IM)
  - Research Site, Savona
  - Research Site, Sora (FR)
  - Research Site, Taormina ME
  - Research Site, Taranto
  - Research Site, Torino
  - Research Site, Viterbo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com